CLINICAL TRIAL: NCT01062919
Title: Postoperative Determinants of Functional Recovery Following Colon Surgery: The Effect of Wound Infiltration With Local Anesthetics
Brief Title: Local Anesthetic Wound Infusion and Functional Recovery After Colon Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate - >70% of colorectal procedures are done laparoscopically
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GEN-08-070
Record Dates: First submitted 2009-09-22; First posted 2010-02-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Colon Cancer; Inflammatory Bowel Diseases; Diverticulitis
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Diverticulitis | interventions — Analgesia, Epidural; Tea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural analgesia group (Experimental): patients in the epidural analgesia group will receive ropivacaine 0.2% through the epidural catheter, normal saline in the wound catheter and PCA with morphine.
  Interventions: Procedure: Epidural analgesia
- Wound Group (Experimental): patients in the epidural analgesia group will receive ropivacaine 0.2% through the wound catheter, normal saline in the epidural catheter and PCA with morphine.
  Interventions: Procedure: Wound catheter

INTERVENTIONS:
Procedure: Epidural analgesia — patients in the epidural analgesia group will receive ropivacaine 0.2% through the epidural catheter, normal saline in the wound catheter and PCA with morphine.
  Other Names: Thoracic epidural analgesia
  Arms: Epidural analgesia group
Procedure: Wound catheter — patients in the epidural analgesia group will receive 0.2%ropivacaine through the wound catheter, normal saline in the epidural catheter and PCA with morphine.
  Other Names: Wound catheter continuous infusion
  Arms: Wound Group

SUMMARY:
This is a double blinded randomized controlled trial in patients undergoing colon open surgery. The purpose is to evaluate the effectiveness of two different analgesic techniques on functional recovery after surgery.

Twenty five patients will receive thoracic epidural analgesia plus patient controlled analgesia (PCA) (epidural analgesia group) and 25 patients wound infiltration of local anesthetic plus PCA (wound infusion group).

Hypothesis: the postoperative recovery of patients receiving local anesthetic wound infusion will be faster than patients receiving thoracic epidural analgesia.

Functional recovery, pain intensity, opioid consumption and side effects, length of hospital stay and biological markers of inflammation after surgery will be measured in both groups.

DETAILED DESCRIPTION:
This is double blinded randomised study of patients undergoing colon open surgery. One group of patients will receive thoracic epidural analgesia plus patient controlled analgesia (PCA) (epidural analgesia group) and the other group will receive infiltration of local anesthetic plus PCA (wound infusion group). Functional restoration, assessed by self-administered quality of Life questionnaires (SF-36, CHAMPS, ICFS) and 2 and 6 min walking test will be assessed in the two groups at 3 and 8 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective open colon surgery

Exclusion Criteria:

* ASA physical status 4
* history of:

  * hepatic failure (liver enzymes abnormally elevated)
  * renal failure (creatinine over 150 mmol/L)
  * cardiac failure
  * organ transplant
  * diabetes
  * morbid obesity (BMI > 40 kg/m-2)
  * chronic use of opioids
  * allergy to local anaesthetics
* History of seizure
* contraindications to the insertion of epidural
* INR > 1.3, PTT > 44 second, platelets < 150.000 per microliter,
* previous spinal surgery limiting the insertion)
* inability to comprehend pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Postoperative functional recovery | at 24, 48, 72 hours, 4 and 8 weeks after the surgery

SECONDARY OUTCOMES:
postoperative pain | at 24, 48, 72 hours after the surgery
opioid consumption | at 24, 48, 72 hours after the surgery
opioid side effects | at 24, 48, 72 hours after the surgery
return of bowel function | at 24, 48, 72 hours after the surgery and continue at the same time everyday until patients have return of bowel function.
length of hospital stay | at 24, 48, 72 hours after the surgery and continue at the same time everyday until the patients are discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, Professor, Principal Investigator — McGill University Healt Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada